CLINICAL TRIAL: NCT06602440
Title: Observations on the Effect of Different Depths of Epidural Catheter Retention on the DPE Technique Combined With the PIEB Mode of Labor Analgesia：a Single-center, Prospective, Randomized Controlled Study
Brief Title: Effect of Epidural Catheter Retention Depth on Labor Analgesia Performed in DPE Combined With PIEB Model
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Peng Liu-2024-2
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Labor Analgesia
Keywords: Uterine contraction pain; Dural puncture epidural technique（DPE）; Programmed intermittent epidural bolus（PIEB）

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3cm group (Other): When performing Dural Puncture Epidural technique with Programmed Intermittent Epidural Bolus（PIEB） mode for labor analgesia, the indwelling depth of the epidural catheter is 3 centimeters.
  Interventions: Procedure: The indwelling length of epidural catheter is 3 centimeters.
- 5cm group (Other): When performing Dural Puncture Epidural technique with Programmed Intermittent Epidural Bolus（PIEB） mode for labor analgesia, the indwelling depth of the epidural catheter is 5 centimeters.
  Interventions: Procedure: The indwelling length of epidural catheter is 5 centimeters.
- 7cm group (Other): When performing Dural Puncture Epidural technique with Programmed Intermittent Epidural Bolus（PIEB） mode for labor analgesia, the indwelling depth of the epidural catheter is 7 centimeters.
  Interventions: Procedure: The indwelling length of epidural catheter is 7 centimeters.

INTERVENTIONS:
Procedure: The indwelling length of epidural catheter is 3 centimeters. — When performing Dural Puncture Epidural technique with Programmed Intermittent Epidural Bolus（PIEB） mode for labor analgesia, According to different indwelling lengths of epidural catheters as variables, patients are divided into three treatment groups（3cm group 、5cm group and 7cm group）
  Arms: 3cm group
Procedure: The indwelling length of epidural catheter is 5 centimeters. — When performing Dural Puncture Epidural technique with Programmed Intermittent Epidural Bolus（PIEB） mode for labor analgesia, According to different indwelling lengths of epidural catheters as variables, patients are divided into three treatment groups（3cm group 、5cm group and 7cm group）
  Arms: 5cm group
Procedure: The indwelling length of epidural catheter is 7 centimeters. — When performing Dural Puncture Epidural technique with Programmed Intermittent Epidural Bolus（PIEB） mode for labor analgesia, According to different indwelling lengths of epidural catheters as variables, patients are divided into three treatment groups（3cm group 、5cm group and 7cm group）
  Arms: 7cm group

SUMMARY:
The purpose of this study is to observe the appropriate indwelling depth of epidural catheter when labor analgesia is performed in the mode of DPE combined with PIEB, and then shorten the onset time of labor analgesia and reduce the occurrence of catheter-related adverse outcomes.

DETAILED DESCRIPTION:
In clinical practice, neuraxial analgesia is the most effective method for labor analgesia, including combined spinal-epidural (CSE) analgesia, dural puncture epidural (DPE) analgesia, and conventional epidural (EP) analgesia. Among them, DPE technology is an improvement of CSE technology. It means using a spinal needle to puncture the dura mater but not injecting drugs into the intrathecal space. Then, the epidural catheter is inserted into the epidural space. The punctured dura mater creates a new pathway for drug displacement from the epidural space to the subarachnoid space. In theory, compared with EP, DPE technology makes drugs enter the subarachnoid space more easily and can achieve a faster onset time of analgesia. At the same time, compared with CSE, the amount of drugs entering the subarachnoid space is not excessive, which can reduce the occurrence of adverse reactions such as itching and hypotension. At present, although there is controversy over the clinical advantages of DPE, its effectiveness has been confirmed in the article published by Gunaydin B et al. in 2019. In a series of RCT trials conducted by Professor Xu Zhendong's team in China, it is believed that the effect of DPE is related to the drug injection mode in the epidural space, the thickness of the puncture needle, and the distance between the drug outlet end and the puncture hole. At the same time, DPE technology combined with programmed intermittent epidural bolus (PIEB) mode seems to be a better choice in labor analgesia. Because the single drug bolus dose generated under the PIEB mode creates greater pressure in the epidural space, which is more conducive to drugs entering the subarachnoid space through the puncture hole. Based on the above research, when performing labor analgesia in the DPE combined with PIEB mode, we believe that the closer the opening of the epidural catheter is to the puncture hole, the easier it is for drugs to generate local pressure around the puncture hole and thus enter the subarachnoid space. This is related to the indwelling depth of the epidural catheter. The shorter the indwelling depth, the more drugs may enter the puncture hole, but it will also increase the probability of catheter detachment. The longer the indwelling depth, the farther the local pressure generated is from the puncture hole, and the advantage of the PIEB mode may be masked. At the same time, an excessively long indwelling depth will increase the incidence of unilateral block.

ELIGIBILITY:
Inclusion Criteria:

1. Those aged 18 to 45 years old;
2. Pregnancy lasts for 37 to 42 weeks;
3. Single healthy pregnant women with cervical dilation < 3.0 cm who wish to use epidural labor analgesia;
4. The NRS score of uterine contraction pain is > 3;
5. ASA grade I-II;
6. BMI ≤ 40 kg/m².

Exclusion Criteria:

1. Those with contraindications to intraspinal anesthesia;
2. Those with a history of allergy to local anesthetics and opioids;
3. Pregnancy diseases (such as pregnancy-induced hypertension, preeclampsia or gestational diabetes, etc.);
4. Known fetal abnormalities or situations associated with an increased risk of cesarean section;
5. Patients who have taken opioids or sedatives within 4 hours before epidural analgesia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Time of satisfactory analgesia. | First dose in the epidural space to NRS score being less than 3.
  The time when the NRS score is less than 3 after the first administration during labor analgesia with DPE combined with PIEB mode.
Consumption of ropivacaine per unit time. | First dose in the epidural space to the end of the third stage of labor.
  The consumption of ropivacaine per unit time during the entire labor analgesia process.

SECONDARY OUTCOMES:
Related adverse outcomes. | First dose in the epidural space to the end of the third stage of labor.
  Occurrence of epidural catheter prolapse, itching, nausea, vomiting, hypotension and unilateral block.
Anesthesia level and lower limb motor block. | When labor analgesia is satisfactory.
  Use the needle prick method to measure the anesthesia level and lower limb motor block after satisfactory labor analgesia.
Duration of labor. | From the onset of labor to its end.
  Duration of the first, second, and third stages of labor.
Changes in fetal heart rate and uterine contraction pressure. | Before and after labor pain.
  Observe the changes in fetal heart rate and uterine contraction pressure before and after labor pain.

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China